CLINICAL TRIAL: NCT04469816
Title: The Family Check-Up for Health: A Family-Centered Health Maintenance Approach to Improve Nutrition and Prevent Obesity in Early Childhood
Brief Title: AFRI Childhood Obesity Prevention Challenge Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FP00008342
Record Dates: First submitted 2020-06-26; First posted 2020-07-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Clinical Trial
Keywords: Hybrid design; Implementation; Effectiveness; Parent Training; Cost-Effectiveness; Primary Care; Integrated Behavioral Health; Family-Based Prevention; Family Check-Up 4 Health; Fidelity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Family Check-Up 4 Health (Experimental): Families will receive the FCU4Health program 3 times annually in a health maintenance model. The FCU4Health coordinator reviews the assessment results with the parents, using motivational interviewing strategies to create a tailored plan to address family needs. This plan may include referrals to community resources or parenting modules that focus on family management.
  Interventions: Behavioral: Family Check-Up 4 Health
- Control-Services as Usual (Experimental): Families will continue with their medical standard of care and referrals for services as appropriate from the healthcare staff in their respective FQHCs or primary healthcare clinics.
  Families will receive brochures about the community programs to which families in the FCU4Health arm are referred.
  Interventions: Other: Services as Usual

INTERVENTIONS:
Behavioral: Family Check-Up 4 Health — A parent-training intervention to improve child health, school readiness and manage obesity.
  Other Names: FCU4Health
  Arms: Behavioral: Family Check-Up 4 Health
Other: Services as Usual — Services/Treatment as usual.
  Arms: Control-Services as Usual

SUMMARY:
This study is a hybrid type 2 effectiveness-implementation trial of the Family Check-Up 4 Health (FCU4Health), an adapted version of the Family Check-Up, in pediatric primary care. Patients will be recruited based on their age (2-5 years old) and randomized to receive the intervention, FCU4Health, or services as usual. All families will be assessed annually over three years.

DETAILED DESCRIPTION:
The FCU4Health is an assessment-driven, Motivational Interviewing (MI) based, parent training program. Parents complete a comprehensive assessment, including questionnaire of the family environment, parenting skills, and child adjustment and health behaviors, and additional observation data. The FCU4Health coordinator reviews the assessment results with the parents, using MI strategies to engage families in making change to support child behavioral health, and to create tailored follow-up services which include parent training modules and referrals to additional support services in the community.

ELIGIBILITY:
Inclusion Criteria:

* Participating caregiver who is at least 18 years of age and understands English and/or Spanish well enough to complete study assessment.

Exclusion Criteria:

* Two exceptions: (1) Children with special needs that preclude engagement in a nutrition-based behavioral intervention (e.g., g-tube dependence) and (2) children who are in state custody.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in the Family Health Behavior Scale | The investigators will examine trajectories of family mealtime routines over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Family Mealtime Routines. Minimum Value: 0. Maximum Value: 20. Where higher scores mean a better outcome.
Changes in the HABITS questionnaire | The investigators will examine trajectories of child food and beverage choices over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Child Food and Beverage Choices. Food Minimum Value: 0. Maximum Value: 24. Where higher food scores mean a better outcome and higher beverage scores mean a worse outcome.
Changes in the Family Health Behavior Scale | The investigators will examine trajectories of child eating behaviors over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Child Eating Behaviors. Minimum Value: 0. Maximum Value: 20. Where higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire | The investigators will examine trajectories of child conduct problems over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Conduct Problems. Minimum Value: 0. Maximum Value: 2. Where higher scores mean a worse outcome.
Children's Behavior Questionnaire | The investigators will examine trajectories of child effortful control over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Effortful Control. Minimum Value: 1. Maximum Value: 5. Where higher scores mean a better outcome.
Strengths and Difficulties Questionnaire | The investigators will examine trajectories of prosocial behavior over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Prosocial Behavior. Minimum Value: 0. Maximum Value: 2. Where higher scores mean a better outcome.
Strengths and Difficulties Questionnaire | The investigators will examine trajectories of emotional problems over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Emotional Problems. Minimum Value: 0. Maximum Value: 2. Where higher scores mean a worse outcome.
Brief Infant Sleep Questionnaire | The investigators will examine trajectories of child sleep routines over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Sleep Routines. Minimum Value: 0. Maximum Value: 24. Where higher scores mean a better outcome.
Media Parenting Scale | The investigators will examine trajectories of child media routines over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Media Routines. Minimum Value: 0. Maximum Value: 24. Where higher scores mean a better outcome.
The Family Health Behavior Scale | The investigators will examine trajectories of child physical activity habits over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Child Physical Activity Habits. Minimum Value: 0. Maximum Value: 24. Where higher scores mean a better outcome.
Trajectories of Community Action for Successful Youth Measure (See Reference Section for citing of title) | The investigators will examine trajectories of parenting warmth over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Parenting Warmth. Minimum Value: 1. Maximum Value: 25. Where higher scores mean a worse outcome.
Trajectories of Community Action for Successful Youth Measure (See Reference Section for citing of title) | The investigators will examine trajectories of family conflict over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Family Conflict. Minimum Value: 0. Maximum Value: 6. Where higher scores mean a worse outcome.
Child-parent relationship scale | The investigators will examine trajectories of parent child conflict over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Parent Child Conflict. Minimum Value: 1. Maximum Value: 25. Where higher scores mean a worse outcome.
Center for Epidemiologic Studies Depression Scale | The investigators will examine trajectories of parent depression over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Depression. Minimum Value: 0. Maximum Value: 80. Where higher scores mean a worse outcome.
Trajectories of Parenting Daily Hassles (See Reference Section for citing of title) | The investigators will examine trajectories of parenting stress over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Parenting Stress. Minimum Value: 1. Maximum Value: 4. Where higher scores mean a worse outcome.
Tool for Substance Use Screening | The investigators will examine trajectories of parent substance use over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Parent Substance Use. Minimum Value: 0. Maximum Value: 1. Where higher scores mean a worse outcome.
Trajectories of Parenting Young Children (See Reference Section for citing of title) | The investigators will examine trajectories of incentive and encouragement over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Incentive and Encouragement. Minimum Value: 0. Maximum Value: 4. Where higher scores mean a better outcome.
Trajectories of Parenting Young Children (See Reference Section for citing of title) | The investigators will examine trajectories of proactive parenting over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Proactive Parenting. Minimum Value: 0. Maximum Value: 4. Where higher scores mean a better outcome.
Trajectories of Parenting Young Children (See Reference Section for citing of title) | The investigators will examine trajectories of parent limit setting over 3 annual assessments (baseline, 1-year, 2-year follow-up).
  Limit Setting. Minimum Value: 0. Maximum Value: 4. Where higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cady Berkel, Ph.D., Principal Investigator — Arizona State University; Justin D. Smith, Ph.D., Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Avondale School District, Avondale, Arizona
  - Bayless Integrated Healthcare, Avondale, Arizona
  - Care1st Avondale Resource and Housing, Avondale, Arizona
  - Arizona State University, Tempe, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crnic KA, Greenberg MT. Minor parenting stresses with young children. Child Dev. 1990 Oct;61(5):1628-37. doi: 10.1111/j.1467-8624.1990.tb02889.x. PMID 2245752
- [Background] McEachern AD, Dishion TJ, Weaver CM, Shaw DS, Wilson MN, Gardner F. Parenting Young Children (PARYC): Validation of a Self-Report Parenting Measure. J Child Fam Stud. 2012 Jun;21(3):498-511. doi: 10.1007/s10826-011-9503-y. PMID 22876108
- [Background] Stormshak EA, DeGarmo D, Garbacz SA, McIntyre LL, Caruthers A. Using Motivational Interviewing to Improve Parenting Skills and Prevent Problem Behavior During the Transition to Kindergarten. Prev Sci. 2021 Aug;22(6):747-757. doi: 10.1007/s11121-020-01102-w. PMID 32036553
- [Derived] Berkel C, Smith JD, Bruening MM, Jordan N, Fu E, Mauricio AM, Grimm KJ, Winslow E, Ray K, Bourne A, Dishion TJ. The Family Check-Up 4 Health: Study protocol of a randomized type II hybrid effectiveness-implementation trial in integrated primary care (the healthy communities 4 healthy students study). Contemp Clin Trials. 2020 Sep;96:106088. doi: 10.1016/j.cct.2020.106088. Epub 2020 Jul 22. PMID 32707101